CLINICAL TRIAL: NCT05543109
Title: Ultrasound Guided Psoas Compartment Block vs Suprainguinal Fascia Iliaca Compartment Block for Pain Management in Pediatric Patients With Developmental Dysplasia Sia of the Hip Joint, Randomized Controlled Trial
Brief Title: Ultrasound Guided Psoas Compartment Block vs Suprainguinal Fascia Iliaca Compartment Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 35635/8/22
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Pain, Postoperative; Hip Dysplasia
MeSH Terms: conditions — Pain, Postoperative; Hip Dislocation | interventions — Fentanyl; Narcotics; Propofol; Anesthetics, Intravenous; Rocuronium; Sevoflurane; Ropivacaine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoas compartment block (Active Comparator): After induction of anesthesia; ultrasound guided psoas compartment block will be done using ropivacaine 0.25% 1ml/kg.
  Interventions: Drug: Fentanyl; Drug: Propofol; Drug: Rocuronium; Drug: Sevoflurane; Drug: Ropivacaine
- Suprainguinal fascia iliaca compartment block (Active Comparator): After induction of anesthesia; ultrasound guided suprainguinal fascia iliaca compartment block will be done using ropivacaine 0.25% 1ml/kg.
  Interventions: Drug: Fentanyl; Drug: Propofol; Drug: Rocuronium; Drug: Sevoflurane; Drug: Ropivacaine

INTERVENTIONS:
Drug: Fentanyl — 1 mic/kg during induction of anesthesia
  Other Names: Narcotic
Drug: Propofol — 3mg/kg during induction of anesthesia
  Other Names: Intravenous anesthetic
Drug: Rocuronium — 0.9 mg/kg during induction of anesthesia
  Other Names: Muscle relaxant
Drug: Sevoflurane — 2-3% during maintanance of anesthesia
  Other Names: Inhalational anesthetic
Drug: Ropivacaine — 0.25% Ropivacaine will be used at 1 ml/kg will be injected Ultrasound guided after induction of general anesthesia.
  Other Names: Local anesthetic

SUMMARY:
The aim of this study was to compare the intraoperative and the postoperative analgesic effect of psoas compartment block (PCB) and supra-inguinal fascia iliaca compartment block (SFIB) in pediatric patients undergoing developmental dysplasia of the hip

DETAILED DESCRIPTION:
All subjects after entering operation room will be connected to standard monitor electrocardiograph, non-invasive blood pressure, heart rate, oxygen saturation.

Three mg/kg of propofol, 0.2 μg/kg of fentanyl and 0.1 mg/kg midazolam will be used for sedation. Oxygen at the concentration of 100% will be administrated under the mask in all patients after satisfactory sedation, tracheal intubation will be performed after intravenous anesthesia with administration of 3 mg/kg of propofol, 0.6 μg/kg of fentanyl and 0.9 mg/kg of rocurium. After intubation 2-3% of sevoflurane and 0.2-0.3 mcg/kg/min of fentanyl will be used to maintain anesthesia guided by PSI and hemodynamic monitoring.

The two groups will receive nerve block with local anesthetics. In the SFIB group, the patients will receive ultrasound-guided SFIB, while the patients in the PCB group will receive PCB under the guidance of ultrasound.

Local anesthetic 0.25% Ropivacaine will be used at 1 ml/kg for SFIB and PCB. (the dose of local anesthetic for SFIB or PCB was not more than 35ml). All blocks will be performed by the same experienced anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing undergo acetabuloplasty
* Anesthesiologists (ASA) physical status of I to II

Exclusion Criteria:

* Known allergy to local anesthetic
* Infection at the block site.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Estimated)
Dates: Start 2022-09-29 (Estimated); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
Intraoperative anesthetic requirement | 1 hour
  Intraoperative anesthetic requirement including intraoperative sevoflurane concentration and total fentanyl consumption
Postoperative analgesic requirements | 8 hours
  Postoperative Ketoprofen and morphine consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Mogahed, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No